CLINICAL TRIAL: NCT00819442
Title: Relationship Between Abnormalities of Desmin Cytoskeleton, Mitochondrial Activity and Expression of Ubiquitin in Aspect of Pathogenesis of Heart Failure and Prognosis.
Acronym: DESMIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Scientific Research and Information Technology, Poland (Other Government)
Collaborators: Polish Academy of Sciences (Other)
Responsible Party: Prof. Robert J. Gil, Polish Academy of Sciences
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: N N402196135
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Dilated Cardiomyopathy
Keywords: heart failure; desmin; ubiquitin
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): patients without heart failure, with cardiobiopsy
  Interventions: Procedure: cardiobiopsy
- 2 (Experimental): patients with heart failure in NYHA class I, II
  Interventions: Procedure: cardiobiopsy
- 3 (Experimental): Patients with heart failure in NYHA class III, IV
  Interventions: Procedure: cardiobiopsy

INTERVENTIONS:
Procedure: cardiobiopsy — 5 samples will be taken from right ventricle by Cordis bioptome

SUMMARY:
The purpose of this study is evaluation of expression of desmin in cardiomyocytes of patients with idiopathic dilated cardiomyopathy. Analysis of relationship between desmin expression and activities of mitochondrium and expression of ubiquitin.

ELIGIBILITY:
Inclusion Criteria:

* idiopatic dilated cardiomyopathy, NYHA I, II, III, IV
* dilated left ventricle
* ejection fraction below 45%

Exclusion Criteria:

* diabetes mellitus
* kidney failure (GFR < 30, creatinine below 2,5 mg/dl

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

SECONDARY OUTCOMES:
qualitative differences in desmin expression in cardiomyocytes of patient with heart failure | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital of Ministry of Internal Affairs and Administration, Warsaw, Poland